CLINICAL TRIAL: NCT01591993
Title: Determination of Sensitive Skin in a Mexican Population by Lactic Acid Testing and Its Analysis Through Biophysical Measures
Brief Title: Determination of Sensitive Skin and Its Biophysical Response in a Latin-American Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Collaborators: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Principal Investigator, Juan Pablo Castanedo Cazares, Dermatology Research Director, Universidad Autonoma de San Luis Potosí
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: SenSk12
Record Dates: First submitted 2012-04-27; First posted 2012-05-04 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Skin Irritancy Tests
Keywords: Sensitive skin; Lactic acid test; Transepidermal water loss; Colorimetry; Capacitance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test subject (Experimental): To each subject, the investigators will randomly apply 10% lactic acid on one nasolabial fold, once.
  Interventions: Procedure: 10% lactic acid test
- Placebo (Placebo Comparator): To each subject, the investigators will apply placebo (0.9% saline solution) on the contralateral nasolabial fold to the lactic acid, simultaneously.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: 10% lactic acid test — To each subject, 10% lactic acid is applied to one nasolabial fold. This will be performed under humidity, temperature and pH control to avoid influence of these variables in the result of the test.
  Arms: Test subject
Procedure: Placebo — To each subject, 0.9% saline solution will be applied to the contralateral nasolabial fold. This will be performed under humidity, temperature and pH control to avoid influence of these variables in the result of the test.
  Arms: Placebo

SUMMARY:
Sensitive skin syndrome is a frequent self-diagnosed entity that has not been previously described in a Latin-american population. One hypothesis to its development is an alteration of the barrier function of the skin. The aim of the study is to describe the frequency of sensitive skin in a mexican population detected through the lactic acid test, and to explore its response through biophysical measures (colorimetry, transepidermal water loss (TEWL) and capacitance). The prevalence of this syndrome in studied populations is approximately 50%. Considering racial skin differences, the investigators would expect at least a 20% prevalence.

For this purpose, the investigators would need a minimum of 243 healthy volunteers, 18 years or older, with previous informed consent, to whom the lactic acid test will be performed. The investigators will record any unpleasant sensation graded in a Visual Analog Scale (VAS) of 10 points, colorimetry, TEWL and capacitance before the test and at 3, 5, 8 and 10 minutes after the lactic acid test.

DETAILED DESCRIPTION:
Sensitive skin is defined as the presence of itching, stinging, burning or other unpleasant sensations due to external factors (such as light, heat, cold, air, cosmetic products, soap, water and even emotional and hormonal factors). By definition it is a subjective syndrome, where there are no clinical signs, making it a self-diagnosed entity. Previous community-based studies, mostly in caucasians, have found a high prevalence in general population. Nonetheless, to date there are only a few studies and with a small amount of subjects that have applied an objective test to identify this syndrome, and even fewer have explored the possible alterations associated to it.

The investigators aim to describe the frequency in a hispanic population, and further explore the presence of alterations in the barrier function through measurement of TEWL and capacitance, as well as possible subclinical erythema (a* axis of colorimetry) or variations due to skin pigmentation (L* axis).

The volunteers in the study will be randomized to receive in one nasolabial fold 10% lactic acid solution, and placebo (0.9% saline solution) in the other to act as the control. The investigators will be grading any unpleasant sensation in a 10-point scale (VAS) at 4 different time intervals: 3, 5, 8 and 10 minutes. The investigators will be measuring colorimetry (ChromaMeter CR-300 (Minolta, Japan)), TEWL (Evaporimeter DermaLab (Cortex Technology, Denmark)) and capacitance (Corneometer DermaLab Moisture Module (Cortex Technology, Denmark)) before performing the test, and at 3, 5, 8 and 10 minutes after it. These time intervals have been previously determined according to previous reports where the maximum intensity of the response is obtained in the first 5 minutes, and after 10 minutes the response gradually diminishes.

Statistical analysis will be performed with square chi test, t-test or U-Mann-Whitney, according to the parametric or non-parametric distribution of the values. All tests will be performed using the JMP software 8.0 (Cary, NC, USA) at 95% of confidence, statistical significance at 5% with 80% power.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Informed consent

Exclusion Criteria:

* Pregnancy
* Known allergy to lactic acid
* Presence of any dermatoses in the nasolabial folds
* Topical o systemic drugs in the previous 4 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2011-10; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Sensitivity to lactic acid | 10 minutes
  Identify and measure the presence of any unpleasant sensation after the application of 10% lactic acid test to the nasolabial fold. Will serve to identify subjects with sensitive skin.

SECONDARY OUTCOMES:
Erythema | 0, 3, 5, 8 and 10 minutes
  Measure the presence of erythema through colorimetry (a* axis).
Skin pigmentation | 0 minutes
  Measure the melanin angle (through L* axis) before performing the test.
Transepidermal water loss | 0, 3, 5, 8 and 10 minutes
  Quantify the change in TEWL by evaporimetry in grams per squared meter per hour, as an indirect measure of skin barrier disfunction.
Capacitance | 0, 3, 5, 8, 10 minutes
  Quantify the change in capacitance by corneometry, as an indirect measure of skin barrier disfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Diana V Hernández-Blanco, MD, Principal Investigator — Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto"; Adriana Ehnis-Pérez, MD, Principal Investigator — Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto"; Juan P Castanedo-Cázares, MD, Study Director — Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto"; Bertha Torres-Álvarez, MD, Study Chair — Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto"
Locations (1):
- Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City, San Luis Potosí, Mexico

REFERENCES:
- [Background] Seidenari S, Francomano M, Mantovani L. Baseline biophysical parameters in subjects with sensitive skin. Contact Dermatitis. 1998 Jun;38(6):311-5. doi: 10.1111/j.1600-0536.1998.tb05764.x. PMID 9687028
- [Background] Issachar N, Gall Y, Borell MT, Poelman MC. pH measurements during lactic acid stinging test in normal and sensitive skin. Contact Dermatitis. 1997 Mar;36(3):152-5. doi: 10.1111/j.1600-0536.1997.tb00399.x. PMID 9145266
- [Background] Sparavigna A, Di Pietro A, Setaro M. 'Healthy skin': significance and results of an Italian study on healthy population with particular regard to 'sensitive' skin. Int J Cosmet Sci. 2005 Dec;27(6):327-31. doi: 10.1111/j.1467-2494.2005.00287.x. PMID 18492170